CLINICAL TRIAL: NCT00987480
Title: A Multicenter Phase II Trial of Hematopoietic Stem Cell Transplantation for the Treatment of Patients With Fanconi Anemia Lacking a Genotypically Identical Donor, Using a Chemotherapy Only Cytoreduction With Busulfan, Cyclophosphamide and Fludarabine
Brief Title: Hematopoietic Stem Cell Transplantation for the Treatment of Patients With Fanconi Anemia Lacking a Genotypically Identical Donor, Using a Chemotherapy Only Cytoreduction With Busulfan, Cyclophosphamide and Fludarabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Boston Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Rockefeller University (Other); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-031; NCT00850317 (obsolete NCT alias); NCT01082133 (obsolete NCT alias)
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Aplastic Anemia; Leukemia; Myelodysplastic Syndrome
Keywords: Stem Cell Transplantation; Anemia; Busulfan; Cyclophosphamide; Fludarabine; 08-031
MeSH Terms: conditions — Anemia, Aplastic; Leukemia; Myelodysplastic Syndromes; Anemia | interventions — Busulfan; fludarabine; Cyclophosphamide; Immunosuppression Therapy; Cyclosporine

ARMS (1):
- chemotherapy-based cytoreductive regimen plus a CD34+ selected (Experimental): This phase II trial is designed to investigate the safety and efficacy of a chemotherapy-based cytoreductive regimen plus a CD34+ selected T-cell depleted peripheral blood stem cell (PBSC) stem cell transplant for the treatment of patients with Fanconi anemia and severe hematologic disease.
  Interventions: Drug: Busulfan, fludarabine, & cyclophosphamide with immunosuppression with ATG and cyclosporine.; Device: CliniMACS device

INTERVENTIONS:
Drug: Busulfan, fludarabine, & cyclophosphamide with immunosuppression with ATG and cyclosporine. — There are three parts in this transplant study. 1) There will be a pre-transplant - preparation - period to see if patient qualifies for the transplant study. This will be done as an outpatient and lasts 2-4 weeks. Once this is completed, there will be 2) the transplant period itself, during which the patient will be admitted and will be an inpatient. This period usually last for 4-6 weeks. Following that, there will be a 3) post transplant period, during which the patient will be watched carefully and monitored in clinic as an out patient. The post transplant period lasts from three months to one year.
Device: CliniMACS device — CD34+ T-cell depleted peripheral blood stem cell transplant

SUMMARY:
This is a genetic disease (transmitted through the parents' genes) called Fanconi Anemia. Because of that genetic disease, the bone marrow has changed and now has failed, or has given rise to a preleukemia called myelodysplastic syndrome (MDS) or leukemia (acute myelogenous leukemia or AML).

Without treatment these complications of Fanconia anemia (FA) are fatal. The only treatment that can cure these complications is an allogeneic transplant of stem cells, meaning, giving the patient bone marrow cells from a healthy donor that can produce normal blood cells that will replace the bone marrow that is sick.

What has been given for the treatment of FA in the past is to use a combination of low doses of radiation to the whole body (total body irradiation) and low doses of the chemotherapy drugs (cyclophosphamide and fludarabine) before the transplant. However, the use of radiation can, later on, increase the chances of getting a second cancer of the skin, head or the neck. These chances of a second cancer are higher than normal in patients with FA.

The purpose of this study is to find out if the doctors can do the same thing with the same chemotherapy drugs used in the past. However physicians will use another chemotherapy drug called busulfan instead of the radiation. The goal of this study is to get rid of the short term and long term risks of the radiation. The first new part of this treatment will be to replace drugs for radiation with chemotherapy drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of Fanconi anemia (confirmed by mitomycin C or diepoxybutane [DEB] chromosomal breakage testing at an approved laboratory).
* Hematologic Diagnosis and Status - Patients must have one of the following hematologic diagnoses:

  * Severe Aplastic Anemia (SAA) with bone marrow cellularity of <25%, or Severe Isolated Single lineage Cytopenia

AND at least one of the following features:

* Platelet count <20 x 109/L or platelet transfusion dependence*
* ANC <1000 x 109/L
* Hgb <8 gm/dl or red cell transfusion dependence*
* Myelodysplastic Syndrome (MDS) (Appendix 1: MDS Classification) - MDS at any stage, based on either one of the following classifications:

  * WHO Classification
  * Refractory anemia and transfusion dependence*
  * Any of other stages
  * IPSS Classification
  * Low risk (score 0) and transfusion dependence*
  * Any other risk groups Score > or = to 0.5
* Acute Myelogenous Leukemia

  * Patients with acute leukemia are included in this trial in remission, refractory or relapsed disease.
  * Transfusion dependence will be defined as greater than ONE transfusion of platelets or red blood cells in the last year prior to evaluation on protocol.

    * Donors:
* Donor choices will be determined by the investigators at each of the centers according to their own institutional criteria.
* All patients evaluated at trial sites and eligible for this trial by virtue of disease and lack of an HLA-genotypically matched related donor will be captured in the database of this trial. Patients who will be enrolled on this protocol must have one of the following donor choices:

  * HLA-compatible Unrelated volunteer donors
  * Patients who do not have a related HLA-matched donor but have an unrelated donor who is either matched at all A, B, C and DRB1 (8/8) loci or who is mismatched at 1/8 loci (A, B, C or DRB1) (7/8) as tested by DNA analysis (high resolution), will be eligible for entry on this protocol.
  * HLA-mismatched Related donors
  * Patients who do not have a related or unrelated HLA-compatible donor must have a healthy family member who is at least HLA-haplotype identical to the recipient. First degree related donors must have a normal DEB test.
  * The donor must be healthy and willing and able to receive a 4-6 day course of G-CSF and undergo 1-3 daily leukaphereses.
  * Related and Unrelated donors must be medically evaluated and fulfill the criteria for collection of PBSCs as per institutional guidelines.

    * Patients:
* Patients and donors may be of either gender or any ethnic background.
* Patients must have a Karnofsky adult, or Lansky pediatric performance scale status > or = 70%.
* At the time of referral for transplantation, patients must have no co-existing medical problems that would significantly increase the risk of the transplant procedure.
* Patients must have adequate physical function measured by :

  * Cardiac: asymptomatic or if symptomatic then 1) LVEF at rest must be > or = to 50% and must improve with exercise or 2) Shortening Fraction > or = to 29%
  * Hepatic: < 5 x ULN SGOT and < 2.0 mg/dl total serum bilirubin.
  * Renal: serum creatinine < or = to 1.5 mg/dl or if serum creatinine is outside the normal range, then CrCl > 60-ml/min/1.73 m2
  * Pulmonary: asymptomatic or if symptomatic, DLCO > 50% of predicted (corrected for hemoglobin)
* Each patient must be willing to participate as a research subject and must sign an informed consent form. Parent or legal guardians of patients who are minors will sign the informed consent form. Assents will be obtained as age appropriate.
* Female patients and donors must not be pregnant or breastfeeding at the time of signing consent. Women must be willing to undergo a pregnancy test prior to transplant and avoid becoming pregnant while on study.

Exclusion Criteria:

* Active CNS leukemic involvement
* Female patients who are pregnant (positive serum or urine HCG) or breast-feeding. Women of childbearing age must avoid becoming pregnant while on study.
* Active uncontrolled viral, bacterial or fungal infection
* Patient seropositive for HIV-I/II; HTLV -I/II

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-09-25 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faird Boulad, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Children's Hospital Boston, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Rockefeller University, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] van Hoogdalem MW, Emoto C, Fukuda T, Mizuno T, Mehta PA, Vinks AA. Population pharmacokinetic modelling of busulfan and the influence of body composition in paediatric Fanconi anaemia patients. Br J Clin Pharmacol. 2020 May;86(5):933-943. doi: 10.1111/bcp.14202. Epub 2020 Jan 23. PMID 31851762
- [Derived] Mehta PA, Davies SM, Leemhuis T, Myers K, Kernan NA, Prockop SE, Scaradavou A, O'Reilly RJ, Williams DA, Lehmann L, Guinan E, Margolis D, Baker KS, Lane A, Boulad F. Radiation-free, alternative-donor HCT for Fanconi anemia patients: results from a prospective multi-institutional study. Blood. 2017 Apr 20;129(16):2308-2315. doi: 10.1182/blood-2016-09-743112. Epub 2017 Feb 8. PMID 28179273
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a multicenter site and MSK is the site responsible for data collection and analysis for all sites.
  11 participants were enrolled at Memorial Sloan Kettering Cancer Center. The remaining 34 participants were enrolled at the participating institutions. This makes a total of 45 participants enrolled and treated on this study.
Period: Overall Study
Arm/Group | Chemotherapy-based Cytoreductive Regimen Plus a CD34+ Selected
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy-based Cytoreductive Regimen Plus a CD34+ Selected
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 8.2 [4.3 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 36
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Successful Neutrophil Engraftment
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy-based Cytoreductive Regimen Plus a CD34+ Selected
Number analyzed (Participants) | 45
Participants
  Achieved neutrophil engraftment | 44
  Did not achieve neutrophil engraftment | 1

2. Primary Outcome: The Incidence of Early Transplant Related Mortality
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy-based Cytoreductive Regimen Plus a CD34+ Selected
Number analyzed (Participants) | 45
Participants | 0

3. Primary Outcome: The Incidence of Acute GvHD
Time Frame: 100 days
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy-based Cytoreductive Regimen Plus a CD34+ Selected
Number analyzed (Participants) | 45
percentage of participants | 6.7

4. Primary Outcome: The Incidence of Chronic GvHD
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy-based Cytoreductive Regimen Plus a CD34+ Selected
Number analyzed (Participants) | 45
Participants
  Developed limited chronic GVHD | 3
  Did not develop limited chronic GVHD | 42

5. Secondary Outcome: Overall Survival at 3 Years
Description: Overall Survival is defined as time from date of transplant to event (death from any cause) or last follow-up.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy-based Cytoreductive Regimen Plus a CD34+ Selected
Number analyzed (Participants) | 45
percentage of participants | 80

6. Secondary Outcome: Disease-free Survival at 3 Years
Description: Defined as time from date of transplant to relapse, graft rejection or graft failure, or death.
  Primary non-engraftment is diagnosed when the participants fails to achieve an ANC >/= 500/ul at any time in the first 28 days post-transplant.
  For participants with MDS or AML, relapse will be analyzed as to type and genetic origin of the MDS/leukemic cells. These will be defined by an increasing number of blasts in the marrow over 5% by the presence of circulating peripheral blasts, or by the presence of blasts in any extramedullary site. Cytogenetic analysis of the marrow and/or peripheral blood will also be obtained for the diagnosis of relapse.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy-based Cytoreductive Regimen Plus a CD34+ Selected
Number analyzed (Participants) | 45
percentage of participants | 77.8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Chemotherapy-based Cytoreductive Regimen Plus a CD34+ Selected
All-Cause Mortality (participants affected / at risk) | 9/45
Serious Adverse Events (participants affected / at risk) | 11/45
Other Adverse Events (participants affected / at risk) | 31/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy-based Cytoreductive Regimen Plus a CD34+ Selected (N=45)
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Blood/Bone Marrow, Other (Blood and lymphatic system disorders) | 1
Cardiopulmonary arrest, cause unknkown (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Death NOS (General disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Gastrointestinal, other (Gastrointestinal disorders) | 1
Hemorrhage, Oral cavity (Gastrointestinal disorders) | 1
Hemorrhage, Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, Stoma (GI) (Gastrointestinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7
Ileus, GI (func obstruction of bowel) (Gastrointestinal disorders) | 1
Inf norm ANC/gr1/2 neut-Blood (Infections and infestations) | 1
Inf norm ANC/gr1/2 neut-Meningitis(meninges) (Infections and infestations) | 1
Inf norm ANC/gr1/2 neut-Myositis infection(muscle) (Infections and infestations) | 1
Infection w/ Gr 3/4 neut, Blood (Infections and infestations) | 1
Infection, other (Infections and infestations) | 4
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 1
Neurology - Other (specify) (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Pneumonitis/pulm infiltrates (Respiratory, thoracic and mediastinal disorders) | 2
Pulm/upp respiratory - Other (spec) (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy-based Cytoreductive Regimen Plus a CD34+ Selected (N=45)
Aspartate aminotransferase increased (Investigations) | 3
Bicarbonate, serum-low (Investigations) | 3
Blood bilirubin increased (Investigations) | 3
Sodium, high (hypernatremia) (Metabolism and nutrition disorders) | 3
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 4
Mucositis (Clin exam)- Pharynx (Gastrointestinal disorders) | 4
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 4
Alanine aminotransferase increased (Investigations) | 5
Infection, other (Infections and infestations) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 6
INR (Investigations) | 6
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 6
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 6
Trglycrde, high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 6
Alkaline phosphatase (Investigations) | 7
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 7
PTT (Investigations) | 7
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 8
Creatinine (Investigations) | 8
Hemoglobin (Investigations) | 8
Hypertension (Vascular disorders) | 8
Leukocytes (total WBC) (Investigations) | 8
Lymphopenia (Blood and lymphatic system disorders) | 8
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 8
Platelets (Investigations) | 8
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 9
AST, SGOT (Investigations) | 10
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 10
ALT, SGPT (Investigations) | 11
Bilirubin (hyperbilirubinemia) (Investigations) | 11
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 14
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT00987480/Prot_SAP_000.pdf